CLINICAL TRIAL: NCT00272402
Title: Reducing Clinical Inertia in Diabetes Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 0308300; R01DK068314 (NIH)
Record Dates: First submitted 2006-01-03; First posted 2006-01-06 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Diabetes Mellitus; Hypertension; Hyperlipidemia
Keywords: physician decision support; diabetes mellitus; electronic medical records; office systems redesign
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Other): Simulated case-based learning
  Interventions: Behavioral: Cognitive Behavioral Intervention
- 2 (Other): EMR clinical decision support tool.
  Interventions: Behavioral: Office System Redesign Intervention
- 3 (No Intervention): Control group

INTERVENTIONS:
Behavioral: Cognitive Behavioral Intervention — Intervention consists of simulated case based learning for physicians.
  Arms: 1
Behavioral: Office System Redesign Intervention — Intervention consists of clinical decision support within the electronic medical record.
  Arms: 2

SUMMARY:
In this randomized trial we evaluate two conceptually distinct but potentially synergistic interventions designed to reduce clinical inertia in the outpatient care of adults with type 2 diabetes. The project addresses the following specific aims;

Specific Aim 1. Implement and assess two conceptually distinct but potentially synergistic interventions to reduce clinical inertia related to control of A1c, SBP, and LDL in adults with diabetes.

* Hypothesis 1. Patients of physicians who receive the Cognitive Behavioral Intervention (CBI) (Group 1) will subsequently have less Clinical Inertia than those who receive no intervention (Group 4).
* Hypothesis 2. Patients of physicians who receive the Office Systems Redesign intervention (CBI) (Group 2) will subsequently have less Clinical Inertia than those who receive no intervention (Group 4).
* Hypothesis 3. Patients of physicians who receive the combined CBI plus OSR intervention (Group 3) will subsequently have less Clinical Inertia than those who receive CBI alone (Group 1) or OSR alone (Group 2).

Specific Aim 2. Assess the impact of interventions to reduce clinical inertia on health care charges.

• Hypothesis 4. After adjustment for baseline measures of health care charges, those who receive no intervention (Group 4), will have higher total health care charges over a 24-month follow-up, relative to the patients of physicians in intervention Group 1, Group 2, or Group 3.

DETAILED DESCRIPTION:
The objective of this project is to improve the care of adults with diabetes (DM) by implementing effective interventions to reduce Clinical Inertia related to control of glycated hemoglobin (A1c), systolic blood pressure (SBP) and LDL-Cholesterol (LDL) in primary care office settings. Clinical inertia is defined as lack of treatment intensification in a patient not at evidence-based goals for A1c, SBP, or LDL. Clinical Inertia (CI) has been implicated as a major factor that contributes to inadequate A1c, SBP, and LDL control, and has been documented in over 80% of primary care office visits in various settings,despite the fact that only 3% to 23% of adults with diabetes have simultaneously achieved A1c < 7%, SBP < 130 mm Hg, and LDL < 100 mg/dl.

In this project we test two interventions designed to reduce clinical inertia. The Cognitive Behavioral Intervention (CBI) is directed at individual primary care physicians and has three components: (a) analyze each physician's clinical moves with diabetes patients to identify patterns that indicate clinical inertia, (b) engage each physician in a series of simulated clinical cases to assess the underlying causes of clinical inertia, and (c) provide each physician with a series of tailored simulated clinical scenarios that are designed to correct the failures of thinking and decision making that result in that physician's observed patterns of clinical inertia. The CBI intervention is based on recent work in cognitive science and learning theory and has been successfully applied in other research and educational settings.

The Office Systems Redesign (OSR) Intervention is also directed to primary care physicians and has three major components: (a) identify specific patients in need of intensified diabetes care and schedule four consecutive monthly office visits with their primary care physician, (b) provide the physician with tailored and specific clinical decision support at the time of each visit based on evidence-based treatment algorithms, (c) implement physician visit resolution and accountability reporting immediately after each visit, using tools adapted from clinical trial protocols.

ELIGIBILITY:
Inclusion Criteria:

Physicians must practice at one of the 18 HPMG clinics and meet all these additional eligibility criteria: (a) be a general internist or family physician, (b) provide ongoing clinical care for 20 or more adults with diabetes mellitus in 2003, and (c) provide written informed consent to participate in the study.

Exclusion Criteria:

None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2006-02; Primary Completion 2008-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Clinical inertia | 12 month post intervention

SECONDARY OUTCOMES:
Direct Medical Costs | 12 month pre and 12 month post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J O'Connor, MD MPH, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Research Foundation, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] O'Connor PJ. Commentary--improving diabetes care by combating clinical inertia. Health Serv Res. 2005 Dec;40(6 Pt 1):1854-61. doi: 10.1111/j.1475-6773.2005.00437.x. No abstract available. PMID 16336552
- [Background] O'Connor PJ, Desai J, Solberg LI, Reger LA, Crain AL, Asche SE, Pearson TL, Clark CK, Rush WA, Cherney LM, Sperl-Hillen JM, Bishop DB. Randomized trial of quality improvement intervention to improve diabetes care in primary care settings. Diabetes Care. 2005 Aug;28(8):1890-7. doi: 10.2337/diacare.28.8.1890. PMID 16043728
- [Result] Sperl-Hillen JM, O'Connor PJ, Rush WA, Johnson PE, Gilmer T, Biltz G, Asche SE, Ekstrom HL. Simulated physician learning program improves glucose control in adults with diabetes. Diabetes Care. 2010 Aug;33(8):1727-33. doi: 10.2337/dc10-0439. PMID 20668151
- [Result] Gilmer TP, O'Connor PJ, Sperl-Hillen JM, Rush WA, Johnson PE, Amundson GH, Asche SE, Ekstrom HL. Cost-effectiveness of an electronic medical record based clinical decision support system. Health Serv Res. 2012 Dec;47(6):2137-58. doi: 10.1111/j.1475-6773.2012.01427.x. Epub 2012 May 11. PMID 22578085
- [Result] O'Connor PJ, Sperl-Hillen JM, Rush WA, Johnson PE, Amundson GH, Asche SE, Ekstrom HL, Gilmer TP. Impact of electronic health record clinical decision support on diabetes care: a randomized trial. Ann Fam Med. 2011 Jan-Feb;9(1):12-21. doi: 10.1370/afm.1196. PMID 21242556